CLINICAL TRIAL: NCT05006326
Title: A Prospective Study of Clinical Application of 68Ga-PSMA PET/MR for Diagnosis and Staging in Hepatocellular Carcinoma
Brief Title: Clinical Application of 68Ga-PSMA PET/MR for Diagnosis and Staging in Hepatocellular Carcinoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Xiaoli Lan, Director of the Department of nuclear medicine, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: XLan-0606-01
Record Dates: First submitted 2021-08-07; First posted 2021-08-16 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2022-02

CONDITIONS: Malignant Neoplasm
MeSH Terms: conditions — Neoplasms | interventions — gallium 68 PSMA-11; Gallium-68; Positron-Emission Tomography; Magnetic Resonance Spectroscopy; Positron Emission Tomography Computed Tomography

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- 68Ga-PSMA PET/MR (Experimental): The investigators selected patients with a high clinical suspicion of HCC, or patients with confirmed HCC without tumour-related treatment who were to be biopsied or surgically resected to obtain pathological results. Patients signed an informed consent form and underwent 68Ga-PSMA PET/MR imaging (or PET/CT imaging if the patient had a contraindication to MR imaging).
  Interventions: Drug: 68Ga-PSMA; Device: PET/MR; Device: PET/CT

INTERVENTIONS:
Drug: 68Ga-PSMA — Intravenous access is established in advance, intravenous bolus injection, 68Ga-PSMA dose is about 1.85-3.7 MBq/kg body weight (0.05-0.1 mCi/kg). Patients were encouraged to drink water after injection and asked to empty their bladder before PET scan.
  Other Names: gallium-68 (68Ga)-prostate specific membrane antigen (PSMA)
Device: PET/MR — Each subject undergoes PET/MR imaging within 40-60 minutes after injection.
  Other Names: Positron Emission Tomography/Magnetic Resonance
Device: PET/CT — Each subject undergoes PET/CT imaging within 40-60 minutes after injection.
  Other Names: Positron Emission Tomography/Computed Tomography

SUMMARY:
In this prospective study, 68Ga-PSMA integrated PET/MR imaging was applied for the diagnosis and staging of hepatocellular carcinoma (HCC). The detection and diagnostic performance of 68Ga-PSMA PET/MR for HCC was evaluated in comparison with the gold standard of puncture biopsy or postoperative pathology. The aim is to make up for the deficiency in FDG PET imaging in the diagnosis and staging of HCC.

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC) is one of the most dangerous malignancies in human health, with the sixth highest incidence of malignant tumors. However, early diagnosis of HCC is difficult. The currently used glucose metabolism imaging agent, 18F-FDG, also accumulates in large amounts in normal liver tissue, which affects the diagnosis of HCC lesions.

Prostate specific membrane antigen (PSMA), a type II transmembrane glycoprotein encoded by the FOLH1 gene, is highly expressed in prostate epithelial cells and has been widely used in the study of prostate cancer. Further studies have found that it is involved in tumor angiogenesis in a variety of solid tumors of non-prostate tissue origin. It is also overexpressed in neovascular endothelial cells of hepatocellular carcinoma, which is significantly associated with tumor grading, staging and prognosis. Moreover, PSMA also has great potential as a target for anti-vascular therapy.

The integrated PET/MR is currently the most advanced imaging device, combining the advantages of PET and MR, with the high sensitivity of PET and the high soft tissue contrast of MR. It has significant advantages over PET/CT in head and neck, abdominopelvic lesions. And MR imaging has no additional radiation and a higher biosafety profile.

In view of the potential of 68Ga-PSMA for HCC imaging, this prospective study proposes to apply 68Ga-PSMA integrated PET/MR imaging for diagnosis and staging of HCC. The detection and diagnostic performance of 68Ga-PSMA PET/MR for HCC was evaluated in comparison with the gold standard of biopsy or postoperative pathology. The aim is to make up for the deficiency in FDG PET imaging in the diagnosis and staging of HCC.

ELIGIBILITY:
Inclusion Criteria:

Each subject must meet all the inclusion criteria to be eligible for the study.

* Subjects or their legal representatives are able to sign an informed consent form
* Subjects are committed to comply with the study procedures and cooperate with the implementation of the full study
* Subjects are 18 years of age or older, regardless of gender
* Subjects with high suspicion of HCC, or diagnosed HCC without tumour-related treatment (supporting evidence including serum AFP, MRI, CT and other imaging data and histopathology), and in good general condition
* Subjects intend to obtain pathological results by biopsy or surgical resection

Exclusion Criteria:

All patients meeting any of the exclusion criteria will be excluded from the study.

* Patients or their legal representatives are unable or unwilling to sign the informed consent form
* Patients are unable to cooperate in the conduct of the full study
* Patients with acute systemic illness and electrolyte disturbances
* Patients with other previous malignancies or a combination of other malignancies
* Patients who are pregnant or lactating women

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-08-16 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and specificity of 68Ga-PSMA PET/MR for diagnosis and staging in hepatocellular carcinoma. | 1 year
  For patients without any treatment, the initial diagnosis and staging results of 68Ga-PSMA PET/MR (PET/CT) will be compared with pathological, clinical and follow-up results.

SECONDARY OUTCOMES:
Correlation of 68Ga-PSMA uptake in HCC patients with PSMA expression levels in tissues. | 1 year
  PSMA-related immunohistochemical staining and quantification of PSMA expression was performed on biopsy/surgical tissue sections from patients. The investigators analysed the correlation between HCC 68Ga-PSMA uptake and PSMA expression levels in tissues.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoli Lan, PhD, Study Director — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Locations (1):
- China, Hubei Province, Wuhan, Hubei, China

REFERENCES:
- [Derived] Qin C, Song X, Sun S, Song Y, Ruan W, Gai Y, Yang M, Wan C, Lan X. [68Ga]Ga-PSMA-617 PET/MRI for imaging patients suspected of hepatocellular carcinoma. Eur J Nucl Med Mol Imaging. 2025 Mar;52(4):1278-1290. doi: 10.1007/s00259-024-06973-7. Epub 2024 Nov 21. PMID 39570398